CLINICAL TRIAL: NCT07238101
Title: Hemodynamic Effects of Fentanyl and Dexmedetomidine in Spine Surgery
Brief Title: Hemodynamic Effects of Fentanyl Vs Dexmedetomidine in Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Ida Julita, dr, Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 216 /KEPK/USU/2024
Record Dates: First submitted 2025-09-23; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Spine Surgery; Hemodynamic Stability During Anesthesia
Keywords: Dexmedetomidine; Fentanyl; Hemodynamics; Anesthesia; Randomized Controlled Trial; Adam Malik Hospital
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Experimental): Participants in this group received dexmedetomidine at a dose of 0.5 μg/kgBW/hour intravenously as part of anesthesia management for spinal surgery. The purpose is to evaluate the effect of dexmedetomidine on hemodynamic stability, including heart rate and mean arterial pressure, during and after induction of anesthesia.
  Interventions: Drug: Dexmedetomidine
- Fentanyl Group (Experimental): Participants in this group received fentanyl at a dose of 1.5 μg/kgBW/hour intravenously as part of anesthesia management for spinal surgery. This arm serves as the comparison group to evaluate differences in hemodynamic parameters such as heart rate and mean arterial pressure compared to dexmedetomidine.
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous administration of dexmedetomidine at a dose of 0.5 μg/kgBW/hour during spinal surgery. Dexmedetomidine is a highly selective alpha-2 adrenergic agonist with sedative and analgesic properties. The aim is to evaluate its effect on maintaining hemodynamic stability, including mean arterial pressure (MAP) and heart rate, during and after anesthesia induction.
  Arms: Dexmedetomidine Group
Drug: fentanyl — Intravenous administration of fentanyl at a dose of 1.5 μg/kgBW/hour during spinal surgery. Fentanyl is a potent synthetic opioid analgesic used to manage pain and modulate hemodynamic responses during surgery. This group serves as the comparator to evaluate differences in hemodynamic parameters, particularly MAP and heart rate, compared to dexmedetomidine.
  Arms: Fentanyl Group

SUMMARY:
Researchers will compare dexmedetomidine to fentanyl to see which drug provides better hemodynamic stability during spinal surgery.

Participants will :

* Receive either dexmedetomidine or fentanyl as part of their anesthesia during elective surgery
* Have their mean arterial pressure and heart rate measured at several time points during the procedure
* Be monitored throughout surgery to assess intraoperative hemodynamic responses and stability

DETAILED DESCRIPTION:
Spinal surgery is frequently associated with perioperative hemodynamic fluctuations and significant postoperative pain. Maintaining stable intraoperative blood pressure and heart rate is essential to minimize surgical bleeding, protect neural structures, and promote optimal recovery. Dexmedetomidine, a highly selective α₂-adrenergic receptor agonist, provides sedation, analgesia, and sympatholytic effects without causing respiratory depression and may contribute to improved cardiovascular stability during anesthesia. Fentanyl, a potent synthetic opioid, is widely utilized as an analgesic adjunct in general anesthesia but may offer less consistent hemodynamic control.

This study is a prospective, interventional, randomized, double-blind controlled trial conducted at Adam Malik General Hospital, Medan, Indonesia, following approval from the institutional ethics committee. A total of 50 adult patients scheduled for elective spinal surgery under general anesthesia were enrolled using consecutive sampling and randomly assigned to receive either dexmedetomidine or fentanyl as part of intraoperative management.

Eligible participants were aged 17-60 years and classified as American Society of Anesthesiologists (ASA) physical status I-III. Patients with known drug hypersensitivity, significant cardiac or vascular abnormalities, or contraindications to the study drugs were excluded.

Hemodynamic parameters, including mean arterial pressure (MAP) and heart rate, were recorded at baseline (T0) and at predetermined intraoperative time points (T1-T12). The primary outcome measure was intraoperative MAP, while secondary outcomes included heart rate and estimated blood loss. Statistical analyses were performed using independent t-tests or Wilcoxon rank-sum tests, with a significance threshold of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 17 and 60 years old
* Classified as ASA physical status 1-3
* Scheduled for elective spinal surgery
* Provided written informed consent

Exclusion Criteria:

* History of drug hipersensitivity to fentanyl or dexmetomidine
* Presence of Cardiac Anatomical abnormalities
* Vsacular disorders or other conditions that may interfere with the study

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Mean Arterial Pressure (MAP) during spinal surgery | MAP will be recorded at baseline (T0), and at 5, 10, 15, 20, 25, 30, 60, 120, 180, and 240 minutes after drug administration
  Measurement of mean arterial pressure (MAP) at multiple time points to compare the effects of dexmedetomidine versus fentanyl on intraoperative hemodynamic stability during spinal surgery.

SECONDARY OUTCOMES:
Change in Heart Rate (Pulse) during spinal surgery | Heart rate will be recorded at the same time points as MAP: baseline (T0), and at 5, 10, 15, 20, 25, 30, 60, 120, 180, and 240 minutes after drug administration
  Measurement of heart rate (pulse) at multiple time points to evaluate hemodynamic response and stability between dexmedetomidine and fentanyl groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Universitas Sumatera Utara, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gilpin B. Changing the public health landscape through advocacy. Circulation. 1997 Apr 15;95(8):1978. doi: 10.1161/01.cir.95.8.1978. No abstract available. PMID 9133498
- [Result] Hasmi. Epidemiological research methods. Jakarta: CV Trans Info Media; 2016.
- [Result] Rizkiya P, Margarita N, Harijono B, Herawati L. Analysis of dexmedetomidine addition in elective major spinal surgery in RSUD Dr. Soetomo. Maj Anestesiol Indones. 2020;9(2):1-9.
- [Result] Yun SH, Song SW, Park JC. Beneficial effects of the addition of intrathecal fentanyl to bupivacaine for spinal anesthesia in cesarean section. Anesth Pain Med (Seoul). 2017;12(3):233-239. doi:10.17085/apm.2017.12.3.233.
- [Result] Park SJ, Shin S, Kim SH, Kim HW, Kim SH, Do HY, Choi YS. Comparison of Dexmedetomidine and Fentanyl as an Adjuvant to Ropivacaine for Postoperative Epidural Analgesia in Pediatric Orthopedic Surgery. Yonsei Med J. 2017 May;58(3):650-657. doi: 10.3349/ymj.2017.58.3.650. PMID 28332374
- [Result] Choi JW, Joo JD, Kim DW, In JH, Kwon SY, Seo K, Han D, Cheon GY, Jung HS. Comparison of an Intraoperative Infusion of Dexmedetomidine, Fentanyl, and Remifentanil on Perioperative Hemodynamics, Sedation Quality, and Postoperative Pain Control. J Korean Med Sci. 2016 Sep;31(9):1485-90. doi: 10.3346/jkms.2016.31.9.1485. PMID 27510395
- [Result] Kaye AD, Chernobylsky DJ, Thakur P, Siddaiah H, Kaye RJ, Eng LK, Harbell MW, Lajaunie J, Cornett EM. Dexmedetomidine in Enhanced Recovery After Surgery (ERAS) Protocols for Postoperative Pain. Curr Pain Headache Rep. 2020 Apr 2;24(5):21. doi: 10.1007/s11916-020-00853-z. PMID 32240402
- [Result] Khosravi F, Sharifi M, Jarineshin H. Comparative Study of Fentanyl vs Dexmedetomidine as Adjuvants to Intrathecal Bupivacaine in Cesarean Section: A Randomized, Double-Blind Clinical Trial. J Pain Res. 2020 Oct 7;13:2475-2482. doi: 10.2147/JPR.S265161. eCollection 2020. PMID 33116789
- [Result] Sahraei R, Ghaedi M, Haghbeen M, Sadegh M, Jahromi S. Comparison of ketamine and dexmedetomidine in reducing complications after laparoscopic cholecystectomy surgery. Med J Islam Repub Iran. 2023;12(2).
- [Result] Emam MWM, Hassan BEDE, Abd El-Hamid HM, Ibrahim IA, Saleh MAE. Comparative study between dexmedetomidine and fentanyl as adjuvants to bupivacaine for postoperative epidural analgesia in abdominal surgery: a randomized controlled trial. Egypt J Anaesth. 2023;39(1):635-641. doi:10.1080/11101849.2023.2238520
- [Result] Sigdel R, Lama M, Gurung S, et al. Intrathecal bupivacaine with fentanyl versus bupivacaine alone in cases undergoing elective cesarean section: comparison of hemodynamics. J Nepal Health Res Counc. 2023;21(2).
- [Result] Hassanin AAM, Ali NS, Elhiny MMMA. Effect of dexmedetomidine versus fentanyl on recovery responses to tracheal extubation in vitrectomy: randomized controlled trial. Egypt J Anaesth. 2023;39(1):40-49. doi:10.1080/11101849.2023.2166617.
- [Result] Ma RX, Qiao RQ, Xu MY, Li RF, Hu YC. Application of Controlled Hypotension During Surgery for Spinal Metastasis. Technol Cancer Res Treat. 2022 Jan-Dec;21:15330338221105718. doi: 10.1177/15330338221105718. PMID 35668701

DOCUMENTS (1):
  • Study Protocol (2025-11-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT07238101/Prot_000.pdf